CLINICAL TRIAL: NCT05340322
Title: Closing the Gap Between Identification and Treatment of Cervical Abnormalities in Lima, Perú Through Integraton of Pocket Colposcopy, Telemedicine and Visual Counseling
Brief Title: Identification and Treatment of Cervical Abnormalities in Perú Through Integration of Pocket Colposcopy and Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00106490
Record Dates: First submitted 2022-04-11; First posted 2022-04-22 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cervical Cancer; HPV Infection; HIV Infections
Keywords: cervical cancer screening; Pap smear; colposcopy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- HPV+ Pap smear (Experimental): Visualization of cervix and if abnormalities are present treat with SOC thermocoagulation.
  Interventions: Device: Colposcopy using pocket colpscope and thermocoagulator

INTERVENTIONS:
Device: Colposcopy using pocket colpscope and thermocoagulator — If HPV+, visualization with pocket colposcope and treatment with thermocoagulator

SUMMARY:
The Pocket colposcope has 510k FDA clearance and has been successfully used in almost 1500 unique patients globally in Duke and non-Duke protocols to date. The objective is to provide colposcopy capability to rural communities in Peru potentially using Telehealth. Approximately 10,000 women will receive self HPV test kit for community health workers. Of these participants, approximately 1,000 HPV+ participants will be invited to participate in this pocket colposcopy study. Approximately 500 of these participants may require treatment using thermocoagulation.

DETAILED DESCRIPTION:
The goal is to demonstrate that the combination of self-sampling, the Pocket colposcope and the thermocoagulator will yield a high proportion of HPV positive women who complete treatment and follow-up care. The bulk of this trial will occur over a two-year period in Peru. Duke will provide the Pocket colposcope and the Calla application to run the device only. Dr. Garcia will recruit and train community women for the distribution of self-collection HPV test kits, identify and partner with 10 to 12 health centers in the Andean region of Peru, conduct baseline data collection in each health center, procure necessary equipment and technology, and conduct training for HPV testing, Pocket colposcopy, and thermocoagulation. Within 18 months trained community women will distribute 10,000 HPV tests to women within the region. The investigators anticipate that 10% of the women screened will be HPV positive and they will be recruited for our trial. As part of the study the participants will be followed to determine if the participants attend a health center, receive Pocket colposcopy, and if needed whether the participants are treated with the thermocoagulator device. All women will be appointed to return to the health center for a follow-up evaluation six months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* HPV+ pap smear
* Women must between the ages of 30-49yo

Exclusion Criteria:

* HPV (-) pap smear
* people without a cervix

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 503 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nimmi Ramanujam, Ph.D., Principal Investigator — Duke University
Locations (1):
- Universidad Peruana Cayetano Heredia, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3734 HPV tests were administered for screening purposes to participate in this study. Of these, 534 women were HPV+. 503 of those were consented to the study
Period: Overall Study
Arm/Group | HPV+ Pap Smear
Started | 503
Completed | 503
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HPV+ Pap Smear
Number analyzed (Participants) | 503
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 503
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 37.49 [30 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 503
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Peru | 503

OUTCOME MEASURES:

1. Primary Outcome: Number of HPV Positive Women Examined
Description: Total number of HPV positive women that went to a Peruvian health center for treatment and were examined using the Pocket Colposcope
Time Frame: up to approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | HPV+ Pap Smear
Number analyzed (Participants) | 503
Participants | 503

2. Secondary Outcome: Number of HPV Positive Women Who Completed the 6 Month Follow-up After Evaluation and Treatment
Time Frame: 6 months after initial visit
Measure: Count of Participants; unit: Participants
Groups:
- HPV+ Pap Smear: Visualization of cervix and if abnormalities are present treat with SOC thermocoagulation.
  Colposcopy using pocket colposcope and thermocoagulator: If HPV+, visualization with pocket colposcope and treatment with thermocoagulator.
Arm/Group | HPV+ Pap Smear
Number analyzed (Participants) | 503
Participants | 488

ADVERSE EVENTS:
Time Frame: Approximately 6 months
Arm/Group | HPV+ Pap Smear
All-Cause Mortality (participants affected / at risk) | 0/503
Serious Adverse Events (participants affected / at risk) | 0/503
Other Adverse Events (participants affected / at risk) | 0/503

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT05340322/Prot_SAP_000.pdf